CLINICAL TRIAL: NCT00557908
Title: The VWD International Prophylaxis (VIP) Study
Brief Title: The Von Willebrand Disease (VWD) International Prophylaxis Study
Acronym: VIP
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Collaborators: Versiti Blood Health (Other); CSL Behring (Industry)
Responsible Party: Principal Investigator, Sharyne M. Donfield, Ph.D., Principal Research Scientist, Skane University Hospital
Other Study IDs: VWD PN
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Von Willebrand Disease
Keywords: Von Willebrand Disease; VWD; prophylaxis
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- VWF/FVIII product infusions: One to three infusions of factor replacement as needed to control bleeding.
  Interventions: Drug: VWF/FVIII products

INTERVENTIONS:
Drug: VWF/FVIII products — Participants in the prospective phase of the study undergo an escalation of treatment from receipt of one to three levels of VWD product. All subjects enrolled will begin treatment on the level one and remain on this regimen for the duration of follow-up, or until they meet the criteria for escalation to level two or three (if indeed they do meet the criteria.)
  Dosing for joint bleeding, epistaxis, and GI bleeding indications: 50 U RCo/kg once per week, 50 U RCo/kg twice per week, or 50 U RCo/kg three times per week.
  Dosing for menorrhagia: 50 U RCo/kg on day 1 of menses for 2 cycles, 50 U RCo/kg on days 1 and 2 of menses for 2 cycles, or 50 U RCo/kg on days 1, 2, and 3 of menses

SUMMARY:
The von Willebrand Disease Prophylaxis Network (VWD PN) is an international study group formed with the goal of investigating the role of prophylaxis in clinically severe VWD that is non-responsive to other treatment(s).

DETAILED DESCRIPTION:
The most common indications for vWD prophylaxis included joint bleeding, epistaxis, gastrointestinal (GI) bleeding, and menorrhagia. Thus, an effort to establish optimal treatment regimens for these indications, through a period of prospective evaluation, is the primary focus of this research. Other goals include a retrospective study of the effect of prophylaxis on bleeding frequency, and a retrospective natural history study of GI bleeding in VWD.

ELIGIBILITY:
Inclusion Criteria:

Type 1: eligible for participation if

* ≤20% RCo and/or ≤20% FVIII; and
* DDAVP non-responsive, defined as occurrence of bleeding episodes not responding satisfactorily to desmopressin, or deemed non-responsive a priori by the investigator; and
* Bleeding indication criteria are met

Type 2: eligible for participation if

* DDAVP non-responsive, defined as occurrence of bleeding episodes not responding satisfactorily to desmopressin, or deemed non-responsive a priori by the investigator; or Type 2B;
* Bleeding indication criteria are met

Type 3: eligible for participation if

* Bleeding indication criteria are met

Bleeding Indication Criteria:

* Joint Bleeding: documentation of at least two apparently spontaneous bleeding episodes in the same joint in the six months prior to enrollment; or three or more apparently spontaneous bleeding episodes in different joints in the six months prior to enrollment.
* GI Bleeding: history of two or more severe GI bleeding episodes associated with either a drop in hemoglobin of ≥ 2 g/dl or requiring red blood cell transfusion or treatment with VWD concentrate.
* Failure to identify other causes of bleeding.
* Menorrhagia: a diagnosis of menorrhagia; prospectively completed Pictorial Blood Assessment Chart score >185 or required treatment with a VWD product for menstrual bleeding on one or more occasions in the year prior to enrollment.
* Normal cervical cytology (PAP) within the six months prior to enrollment for females ≥ 18 years of age.
* Epistaxis 1. Three or more bleeding episodes in a six-month period that required treatment with VWD concentrates or red cell transfusions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The VWD population includes those with Type 1 if </=20% RCo and/or </=20% FVIII; and DDAVP non-responsive; Type 2 if DDAVP non-responsive, or Type 2B; and Type 3; who meet bleeding indication criteria having defined patterns of gastrointestinal bleeding, joint bleeding, epistaxis, or menorrhagia.
  Individuals already on prophylaxis for VWD, for any indication, and individuals who were on a regimen of prophylaxis for at least six months that was discontinued because it was no longer required, or those with a history of GI bleeding due either to proven angiodysplasia or unexplained by other factors.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2007-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
von Willebrand Disease associated bleeding frequency | 1 year

SECONDARY OUTCOMES:
Optimal treatment regimens for joint bleeding, GI bleeding, epistaxis, and menorrhagia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Erik Berntorp, MD, PhD, Principal Investigator — Skåne University Hospital, Malmö, Sweden; Thomas Abshire, MD, Principal Investigator — Versiti Blood Health
Locations (3):
- United States (2):
  - Rho, Inc., Chapel Hill, North Carolina
  - BloodCenter of Wisconsin, Milwaukee, Wisconsin
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Holm E, Abshire TC, Bowen J, Alvarez MT, Bolton-Maggs P, Carcao M, Federici AB, Gill JC, Halimeh S, Kempton C, Key NS, Kouides P, Lail A, Landorph A, Leebeek F, Makris M, Mannucci P, Mauser-Bunschoten EP, Nugent D, Valentino LA, Winikoff R, Berntorp E. Changes in bleeding patterns in von Willebrand disease after institution of long-term replacement therapy: results from the von Willebrand Disease Prophylaxis Network. Blood Coagul Fibrinolysis. 2015 Jun;26(4):383-8. doi: 10.1097/MBC.0000000000000257. PMID 25688461
- [Result] Makris M, Federici AB, Mannucci PM, Bolton-Maggs PHB, Yee TT, Abshire T, Berntorp E. The natural history of occult or angiodysplastic gastrointestinal bleeding in von Willebrand disease. Haemophilia. 2015 May;21(3):338-342. doi: 10.1111/hae.12571. Epub 2014 Nov 7. PMID 25381842
- [Result] Abshire TC, Federici AB, Alvarez MT, Bowen J, Carcao MD, Cox Gill J, Key NS, Kouides PA, Kurnik K, Lail AE, Leebeek FW, Makris M, Mannucci PM, Winikoff R, Berntorp E; VWD PN. Prophylaxis in severe forms of von Willebrand's disease: results from the von Willebrand Disease Prophylaxis Network (VWD PN). Haemophilia. 2013 Jan;19(1):76-81. doi: 10.1111/j.1365-2516.2012.02916.x. Epub 2012 Jul 23. PMID 22823000
- [Result] Berntorp E, Abshire T; von Willebrand Disease Prophylaxis Network Steering Committee. The von Willebrand disease prophylaxis network: exploring a treatment concept. J Thromb Haemost. 2006 Nov;4(11):2511-2. doi: 10.1111/j.1538-7836.2006.02179.x. No abstract available. PMID 17059476